CLINICAL TRIAL: NCT01056328
Title: Irrigated Ablation System Evaluation for AF
Brief Title: Irrigated Ablation System Evaluation for Atrial Fibrillation (AF)
Acronym: IRASE-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 90030928
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- St. Jude Medical Cardiac Ablation System (Experimental)
  Interventions: Device: SJM Irrigated Cardiac Ablation System
- FDA approved Open Irrigated Radio Frequency Ablation System (Active Comparator)
  Interventions: Device: FDA approved Open Irrigated RF Ablation System

INTERVENTIONS:
Device: SJM Irrigated Cardiac Ablation System — Irrigated ablation catheter
  Arms: St. Jude Medical Cardiac Ablation System
Device: FDA approved Open Irrigated RF Ablation System — Irrigated ablation catheter
  Arms: FDA approved Open Irrigated Radio Frequency Ablation System

SUMMARY:
The purpose of this study is to test the safety and effectiveness of an Irrigated Ablation System for the treatment of symptomatic paroxysmal atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Signed Patient Informed Consent Form
* Able and willing to comply with all pre-, post-, and follow-up testing and requirements
* Failure of at least one anti-arrhythmic medication (AAD) for paroxysmal atrial fibrillation* [class I or III, or AV nodal blocking agents such as beta blockers (BB) and calcium channel blockers (CCB)] as evidenced by recurrent symptomatic paroxysmal atrial fibrillation*, or intolerable side effects due to AAD
* Subjects with symptomatic paroxysmal atrial fibrillation (PAF)*

  * PAF is defined as recurrent atrial fibrillation (AF) that terminates spontaneously within seven days.

Exclusion Criteria:

* Atrial fibrillation (AF) secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause
* Previous ablation for AF
* History of any valvular cardiac surgical procedure
* Coronary artery bypass grafting (CABG) procedure within the last six months
* Awaiting cardiac transplantation or other cardiac surgery within the next 12 months
* Left atrial thrombus
* History of a documented thromboembolic event within the past one (1) year
* Diagnosed atrial myxoma
* An implanted implantable cardioverter defibrillator (ICD)
* Significant pulmonary disease, (e.g. restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces chronic symptoms
* Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study
* Women who are pregnant (by history of menstrual period or pregnancy test if the history is considered unreliable)
* Acute illness or active systemic infection or sepsis
* Unstable angina
* Myocardial infarction within the previous two months
* Left ventricular ejection fraction (LVEF) <40% as determined by pre-procedure transthoracic echocardiogram (TTE)
* History of blood clotting or bleeding abnormalities
* Contraindication to anticoagulation (i.e. heparin or warfarin)
* Contraindication to computed tomography/magnetic resonance angiography (CT/MRA) procedure
* Life expectancy less than 12 months
* Enrollment in an investigational study evaluating another device or drug
* Uncontrolled heart failure or New York Heart Association (NYHA) class III or IV heart failure
* An intramural thrombus tumor, or other abnormality that precludes catheter introduction or manipulation
* Presence of a condition that precludes vascular access
* Left atrial size ≥ 50 mm as determined by pre-procedure TTE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2010-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (27):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Arrhythmia Consultants/Scottsdale Healthcare, Scottsdale, Arizona
  - Good Samaritan Hospital, Los Angeles, California
  - University of Californai, San Diego Medical Center, San Diego, California
  - Colorado Cardiac Alliance, Colorado Springs, Colorado
  - Diagnostic Cardiology Associates, P.A.; St. Vincents Medical Center, Jacksonville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University Hospital, Midtown, Emory, Georgia
  - University of Kansas Hospital, Kansas City, Kansas
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Spectrum Health, Grand Rapids, Michigan
  - MAHI, Saint Luke's Hospital, Kansas City, Missouri
  - NYU Langone Medical Center, New York, New York
  - Mount Sinai Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Centennial Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Baylor Heart & Vascular Hospital, Dallas, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - Intermountain Medical Center, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Inova Fairfax Hospital / Inova Heart and Vascular Institute, Falls Church, Virginia
- Sunybrook Health Sciences Centre, Toronto, Ontario, Canada
- South Korea (2):
  - Severance Hospital, Seoul
  - Korea University Anam Hospital, Seoul

RESULTS

PARTICIPANT FLOW:
Groups:
- SJM Cardiac Ablation System: SJM Irrigated Cardiac Ablation System: Irrigated ablation catheter
- FDA Approved Open Irriagated RF Ablation System: FDA approved Open Irrigated RF Ablation System: Irrigated ablation catheter
Period: Overall Study
Arm/Group | SJM Cardiac Ablation System | FDA Approved Open Irriagated RF Ablation System
Started | 164 | 160
Completed | 147 | 144
Not Completed | 17 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SJM Cardiac Ablation System | FDA Approved Open Irriagated RF Ablation System | Total
Number analyzed (Participants) | 164 | 160 | 324
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (12.4) | 60.6 (9.7) | 59.5 (11.2)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 96 | 96 | 192
  >=65 years | 68 | 64 | 132
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 66 | 125
  Male | 105 | 94 | 199
Region of Enrollment [Number; unit: participants]
  United States | 149 | 149 | 298
  Korea, Republic of | 9 | 7 | 16
  Canada | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Confirmation of Entrance Block in the Pulmonary Veins
Time Frame: 20 minutes after initial isolation
Measure: Number; unit: participants
Arm/Group | SJM Cardiac Ablation System | FDA Approved Open Irriagated RF Ablation System
Number analyzed (Participants) | 164 | 160
participants | 159 | 157

2. Primary Outcome: Incidence of Adverse Events Included in the Pre-specified Composite
Description: Atrial perforation, atrio-esophageal fistula, cardiac tamponade, cerebrovascular accident, death, diaphragmatic paralysis, hospitalization, myocardial infarction, pericaridal effusion, pericarditis, pulumonary edema, pulmonary vein stenosis, thromboembolism, transient ischemic attack, and vascular access complications.
Time Frame: 7 days
Measure: Number; unit: participants
Groups:
- St Jude Medical (SJM) Cardiac Ablation System: SJM Irrigated Cardiac Ablation System: Irrigated ablation catheter
- FDA Approved Open Irrigated RF Ablation System: FDA approved Open Irrigated Radio Frequency (RF) Ablation System: Irrigated ablation catheter
Arm/Group | St Jude Medical (SJM) Cardiac Ablation System | FDA Approved Open Irrigated RF Ablation System
Number analyzed (Participants) | 134 | 131
participants | 7 | 6

3. Primary Outcome: Incidence of Adverse Events Included in the Pre-specified Composite.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | SJM Cardiac Ablation System | FDA Approved Open Irriagated RF Ablation System
Number analyzed (Participants) | 134 | 131
participants | 12 | 13

4. Secondary Outcome: Documented (> 30 Seconds) Asymptomatic Episodes of Atrial Fibrillation (AF), Atrial Flutter (AFL), or Atrial Tachicardia (AT) After the Blanking Period
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | SJM Cardiac Ablation System | FDA Approved Open Irrigated RF Ablation System
Number analyzed (Participants) | 147 | 131
participants | 116 | 119

5. Secondary Outcome: Early Onset (Within 90 Days) of SAE/Non-serious AEs and Late Onset (After 90 Days) SAEs
Description: Early onset (within 90 days) of Serious Adverse Events (SAE)/Non-serious Adverse Events (AEs) and late onset (after 90 days) Serious Adverse Events (SAEs)
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | SJM Cardiac Ablation System | FDA Approved Open Irriagated RF Ablation System
Number analyzed (Participants) | 158 | 157
participants | 40 | 26

ADVERSE EVENTS:
Arm/Group | SJM Cardiac Ablation System | FDA Approved Open Irrigated RF Ablation System
Serious Adverse Events (participants affected / at risk) | 26/164 | 16/160
Other Adverse Events (participants affected / at risk) | 14/164 | 10/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SJM Cardiac Ablation System (N=164) | FDA Approved Open Irrigated RF Ablation System (N=160)
Pulmonary vein stenosis (Cardiac disorders) | 5 (5) | 7 (7)
Cardiac perforation (Cardiac disorders) | 1 (1) | 1 (1)
Chest and back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 2 (2) | 0 (0)
Local hematoma (Vascular disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery spasm (Cardiac disorders) | 0 (0) | 2 (2)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Other (General disorders) | 8 (8) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SJM Cardiac Ablation System (N=164) | FDA Approved Open Irrigated RF Ablation System (N=160)
Chest and back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Local hematoma (Vascular disorders) | 3 (3) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pseudoaneurysm (Vascular disorders) | 0 (0) | 1 (1)
Skin burn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Other (General disorders) | 6 (6) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other